CLINICAL TRIAL: NCT06018415
Title: Effects of Early and Late Time-restricted Eating on Overweight Adults With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.XJTU1AF2023LSK-398
Record Dates: First submitted 2023-08-13; First posted 2023-08-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Syndrome; Overweight and Obesity; Time Restricted Eating
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early time-restricted eating (eTRE) (Experimental): The eTRE group is instructed to consume all calories from 7 AM to 3 PM each day and fast from 3 PM to 7 AM
  Interventions: Behavioral: Early time-restricted eating (eTRE)
- Late time-restricted eating (lTRE) (Experimental): The lTRE group is instructed toconsume all calories from 11 AM to 7 PM each day and fast from 7 PM to 11 PM
  Interventions: Behavioral: Late time-restricted eating (lTRE)

INTERVENTIONS:
Behavioral: Early time-restricted eating (eTRE) — The eTRE group is instructed to consume all calories in early 8h eating window,
  Arms: Early time-restricted eating (eTRE)
Behavioral: Late time-restricted eating (lTRE) — The lTRE group is instructed to consume all calories in late 8h eating window.
  Arms: Late time-restricted eating (lTRE)

SUMMARY:
Investigators aim to compare the effects of early and late time-restricted feeding on overweight adults with metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years
2. Body mass index (BMI): 24.0-40.0 kg/m2
3. Diagnosed with metabolic syndrome (i.e., more than 3 abnormal findings out of 5):

   1. Waist circumference ≥ 90 cm (men) or ≥ 80 cm (women).
   2. Elevated triglyceride (TG) (use of lipid-lowering medication is an alternate indicator) ≥ 150 mg/dL (1.7 mmol/L).
   3. Reduced high-density lipoprotein cholesterol (HDL-c) (use of lipid-lowering medication is an alternate indicator) < 40 mg/dL (1.0 mmol/L) in males < 50 mg/dL (1.3 mmol/L) in females.
   4. Elevated blood pressure (use of antihypertensive medication is an alternate indicator). Systolic blood pressure (SBP) ≥ 130 and/or diastolic blood pressure (DBP) ≥ 85 mmHg.
   5. Elevated fasting blood glucose (FBG) (used of hypoglycemic medications is an alternate indicator) ≥ 100 mg/dL (5.6 mmol/L).

Exclusion Criteria:

1. Unstable weight (change > 10% current body weight) for 3 months prior to the study
2. Pregnant or breast-feeding
3. Night shift workers
4. History of major diseases or related diseases, such as cancer, inflammatory disease, chronic obstructive pulmonary disease and major adverse cardiovascular event
5. Active viral hepatitis, acquired immune deficiency syndrome, syphilis and other sexually transmitted diseases, tuberculosis and other infectious diseases
6. Being treated with antibiotics or corticosteroids
7. Current participate in other weight-management program, current on a prescribed diet for special disease or current on any drugs that effect appetite
8. The researcher deemed it inappropriate to participate in the experimenter.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | 0-week; 6-week and 12-week
  Body weight is assessed at the research center with the participants without shoes and in light clothing using a digital scale (OMRON MEDICAL Beijing Co., Ltd. HNH-318) to the nearest 0.1 kg.
Changes in abdominal fat area | 0-week; 6-week and 12-week
  Abdominal fat area is measured using bioelectrical impedance analysis (OMRON MEDICAL Beijing Co., Ltd. DUALSCAN, HDS-2000) to the nearest 1 cm2.

SECONDARY OUTCOMES:
Changes in body composition ( body fat mass) | 0-week and 12-week
  Body composition (body fat mass ) is measured using the dual-energy X-ray absorptiometry (DXA, Hologic Serie horzion-wi QDR., Bedford, MA, USA)
Changes in body composition (body muscle mass) | 0-week and 12-week
  Body composition ( body muscle mass) is measured using the dual-energy X-ray absorptiometry (DXA, Hologic Serie horzion-wi QDR., Bedford, MA, USA)
Changes in glycemic control | 0-week; 6-week and 12-week (glucose and insulin)0-week and 12-week (HbA1c)
  Plasma glucose is measured on an automatic biochemistry analyzer (HITACHI, Inc.; LAbOSPECT, 008AS) using standard reagents to the nearest 0.01 mmol/L; Serum insulin is measured by a magnetic particle chemiluminescence immunoassay (Kaeser 6600, Guangzhou Kangrun Co., Ltd., China) to the nearest 0.01 μIU/mL;
Changes in hemoglobin A1c (HbA1c) | 0-week; 6-week and 12-week (glucose and insulin)0-week and 12-week (HbA1c)
  HbA1c is measured on an automatic HbA1c analyzer (TOSOH BIOSCIENCE, Inc.; HLC-723G8) to the nearest 0.1%.
Changes in total cholesterol, triglyceride (TG), high-density lipoprotein cholesterol (HDL-c), and low-density lipoprotein cholesterol (LDL-c) | 0-week; 6-week and 12-week
  Plasma lipids of total cholesterol, TG, HDL-c, and LDL-c are measured on an automatic biochemistry analyzer (HITACHI, Inc.; LAbOSPECT, 008AS) using standard reagents to the nearest 0.01 mmol/L.
Changes in uric acid (UA) | 0-week; 6-week and 12-week
  UA is measured on an automatic biochemistry analyzer (HITACHI, Inc.; LAbOSPECT, 008AS) using standard reagents to the nearest 1 µmol/L.
Changes in blood pressure. | 0-week; 6-week and 12-week
  Blood pressure is measured in triplicate using a digital automatic blood pressure (Omron HBP-9020, Kyoto, Japan) to the nearest 1 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Bingyin Shi, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.